CLINICAL TRIAL: NCT01953809
Title: A Phase 1, Randomized, Single Blind Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of an Oral Contraceptive Containing Norethindrone and Ethinyl Estradiol When Co-administered With GSK1322322 in Healthy Adult Women of Childbearing Age Who Are of Non-Childbearing Potential Due to Surgical Sterilization or IUD Placement (PDF112163)
Brief Title: A Pharmacokinetics, Pharmacodynamics, and Safety Study of an Oral Contraceptive Containing Norethindrone and Ethinyl Estradiol When Co-administered With GSK1322322 in Healthy Adult Women
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Emerging GSK1322322 pre-clinical data ID'd potentially reactive metabolites previously not seen that changed the risk: benefit profile and led to a termination
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 112163
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Infections, Bacterial
Keywords: oral; oral contraceptive; pharmacokinetics; drug interaction; pharmacodynamics; GSK1322322; antibiotic; safety
MeSH Terms: conditions — Bacterial Infections | interventions — GSK1322322

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Run-in Period (Experimental): All subjects will receive EE/NE for first 21 days and EE/NE matching placebo for next 7 days before start of treatment phase
  Interventions: Drug: EE/NE; Drug: EE/NE Placebo
- Group 1 (Experimental): Subjects upon completion of 28 days of run-in period will receive GSK1322322/Placebo + EE/NE in period 1 and only EE/NE in period 2 and 3 of treatment phase. Each period will be of 7 days
  Interventions: Drug: GSK1322322; Drug: EE/NE; Drug: GSK1322322 Placebo
- Group 2 (Experimental): Subjects upon completion of 28 days of run-in period will receive only EE/NE in period 1, GSK1322322/Placebo + EE/NE in period 2 and again EE/NE only in period 3 of treatment phase. Each period will be of 7 days
  Interventions: Drug: GSK1322322; Drug: EE/NE; Drug: GSK1322322 Placebo
- Group 3 (Experimental): Subjects upon completion of 28 days of run-in period will receive only OC in period 1 and 2, and GSK1322322/Placebo + EE/NE in period 3 of treatment phase. Each period will be of 7 days
  Interventions: Drug: GSK1322322; Drug: EE/NE; Drug: GSK1322322 Placebo

INTERVENTIONS:
Drug: GSK1322322 — Oral tablets with unit dose strength of 500mg and dose level of 1500mg (3 x 500mg) for twice a day administration for 7 days in treatment phase
  Arms: Group 1; Group 2; Group 3
Drug: EE/NE — Oral contraceptive tablet containing 0.035mg EE and 1mg NE for once daily administration for 21 days in run-in phase and 21 days in treatment phase
Drug: GSK1322322 Placebo — GSK1322322 matching placebo tablets for twice a day administration (3 tablets each time) for 7 days in treatment period.
  Arms: Group 1; Group 2; Group 3
Drug: EE/NE Placebo — EE/NE matching placebo tablet for once daily administration for 7 days in run-in phase.
  Arms: Run-in Period

SUMMARY:
This study is being conducted to confirm that GSK1322322 has no negative impact on hormone levels and contraceptive efficacy when co-administered with a frequently prescribed oral contraceptive thereby to facilitate the use of GSK1322322 in women of child-bearing potential receiving oral contraceptive (OC) pre-infection. This study is designed to investigate steady-state plasma ethinyl estradiol (EE) and norethindrone (NE) pharmacokinetic (PK) following administration of Ortho-Novum (EE/NE) 1 tablet every 24 hours (q24h) fed with and without GSK1322322 1500 milligram (mg) q12h fed. Each subject will participate in the study for approximately 12 weeks: a 30 day screening period, 4-week run-in period, three 7 day treatment periods, and a 3-5 day follow-up period. The study is planned to enroll approximately 24 subjects (18 active/6 placebo).

DETAILED DESCRIPTION:
Please note that Ortho-Novum is a registered trademark of Ortho Pharmaceutical Corporation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator feels that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Non smoking female (of childbearing age), between 18 and 45 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy without oophorectomy (at least one functioning ovary required) or child bearing age with the presence of non-drug eluting intra uterine device (IUD) i.e. copper. NOTE: The IUD placement needs to be confirmed by an obstetrician-gynecologist.
* Subjects must be willing to use EE/NE in combination with one of the following appropriate contraceptive methods from at least 14 days prior to the first dose of study drug until completion of the follow-up visit Complete abstinence from intercourse for at least 14 days prior to the first dose of IP, throughout the study, and for the subsequent post study monitoring or; A barrier method plus a spermicide (e.g., condom or diaphragm with spermicidal foam/gel/cream/ suppository for at least 14 days prior to the first dose of IP throughout the study, and for the subsequent post study monitoring or Sterilization (vasectomy) of male partner prior to commencement of female subject's last normal menstrual period prior to IP administration and the male partner is the sole partner for that female subject
* Body weight >=50 kilograms (kg) (110 pounds [lbs]) and <114kg (<250 lbs) and body mass index within the range 19 to 32 kg/meter^2 (inclusive).
* Alanine aminotransferase, alkaline phosphatase and bilirubin <=1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening and check-in (repeat allowed at check-in only).
* QT interval corrected for heart rate by Bazett's formula (QTcB) < 450 millisecond (msec) at screening and check-in.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* Pregnant females as determined by positive human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* History of any condition that would contraindicate Ortho-Novum administration (including hypertension, stroke, ischemic heart disease, venous thromboembolism or family history of thromboembolism, known factor V Leiden mutation or other gene mutations associated with increased risk of thromboembolism, migraine headaches, carcinoma of the breast, liver or endometrium, gallbladder disease, history of undiagnosed abnormal uterine bleeding, etc.
* Females with conditions or concurrent medications that could adversely affect hormone levels (e.g. oophorectomies).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Endocrine system: untreated or unstable thyroid disorder and/or diabetes mellitus (I and II). Treatment of the condition must be stable for at least 4 weeks prior to first dose of study drug.
* Have suffered a urinary tract, bladder, or vaginal infection within 4 weeks prior to the first dose of study drug, or has a urinalysis result at Screening consistent with an urinary tract infection. Subjects diagnosed with an infection at Screening should be treated appropriately and may be re-screened after 4 weeks.
* Fasting triglycerides > 300 mg/deciliter (dL) at Screening.
* A positive pre-study Hepatitis B surface antigen, positive Hepatitis C antibody, or a positive test for human immuno virus (HIV) antibody result within 3 months of screening.
* A positive pre-study drug/alcohol screen.
* History of regular alcohol consumption within 6 months of the study defined as An average weekly intake of >7 drinks for females. One drink is equivalent to 12 gram of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Concurrent-medications that alter gastro-intestinal motility result in diarrhea or bind study drugs (for example erythromycin, antacids, prokinetic agents, cholestyramine).
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety due to potential drug interaction.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or regular use of tobacco- or nicotine-containing products within 4 weeks prior to screening.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices] from 7 days prior to the first dose of study medication.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination):

Female subjects with Heart rate <50 and >100 beats per minute (bpm), PR interval <120 and >220 msec, QRS duration <70 and >120 msec, QTcB >=450 msec (Note: The waveforms must enable the QT interval to be clearly defined), Q wave>30 msec Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization).

Any conduction abnormality (including but not specific to left or right bundle branch block, AV block (2nd degree or higher), Wolf Parkinson White (WPW) syndrome), sinus pauses> 3 seconds, non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual subject.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Composite of PK parameters of EE/NE to compare the steady state plasma PK. If data permit, after EE/NE alone for 7 days and after EE/NE with GSK1322322 for 7 days. | Plasma PK samples will be collected at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours on Day 7, 14 and 21 of both run-in phase and on treatment phase.
  PK parameters include: steady-state area under the concentration-time curve over the dosing interval (AUC[0-tau]), maximum observed concentration (Cmax), time of occurrence of Cmax (Tmax), minimum observed concentration (Cmin), and terminal phase half-life (t1/2)

SECONDARY OUTCOMES:
Composite of PK parameters of GSK1322322 following co-administration of GSK1322322 and EE/NE for 7 days | Plasma PK samples will be collected at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hours post morning dose on day 7, 14, and 21 of treatment phase.
  PK parameters include: steady-state AUC(0-tau), Cmax, Tmax
Number of subjects with adverse events (AEs) as a measure of safety and tolerability | 8 weeks
  AEs will be collected from the start of Study Treatment and until the follow-up contact.
Concurrent medication assessment as a measure of safety and tolerability | 8 weeks
Laboratory parameter assessment as a measure of safety and tolerability | 8 weeks
  Laboratory parameters include: hematology, clinical chemistry, urinalysis and additional parameters
Electrocardiogram (ECG) assessment as a measure of safety and tolerability. | 8 weeks
  12-lead ECGs will be obtained at each time point using an ECG machine that automatically to calculate the heart rate and measures PR, QRS, QT, and QT interval corrected for heart rate
Vital sign measurement as a measure of safety and tolerability | 8 weeks
  Vital sign measurements will include systolic and diastolic blood pressure, temperature, and pulse rate
Pre-dose serum level of Lutenizing Hormone (LH). | 7 weeks
  LH will be evaluated as surrogate marker of contraceptive efficacy
Pre-dose serum level of Follicle stimulating hormone (FSH) | 7 weeks
  FSH will be evaluated as surrogate marker of contraceptive efficacy
Pre-dose serum level of Progesterone | 7 weeks
  Progesterone will be evaluated as surrogate marker of contraceptive efficacy

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline